CLINICAL TRIAL: NCT06264765
Title: Comparison Of The Effect Of Scalp Block And Incision Sıte Infiltratıon Applied On Postoperative Acute Paın And Hemodynamics In Patients Undergoing Craniotomy
Brief Title: Scalp Block -Craniotomi
Acronym: scalp block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, ANESTHESİOLOGİST, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 22-12-23
Record Dates: First submitted 2023-12-22; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hemodynamic Instability
Keywords: scalp block; opioid consumption; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized double blinding
Who Masked: Participant, Care Provider
Masking Description: Blind patients and postoperative follow-ups will not know which group the patient is in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scalp block (Other): Following induction of anesthesia, a scalp block will be performed before the surgery begins.
  Interventions: Other: scalp block
- incisional infiltration (Other): Following induction of anesthesia, incisional infiltration will be performed before the surgery begins.
  Interventions: Other: Incisional infiltration

INTERVENTIONS:
Other: scalp block — The scalp block will be performed by the anesthesiologist 10 minutes before the pin head holder application (PHHA). Supraorbital and supratrochlear nerves will be blocked bilaterally with 6 ml of 0.5% bupivacaine injected vertically into the skin above the eyebrow midline. Auriculotemporal nerves will be blocked bilaterally by injecting 4 ml of 0.5% bupivacaine 1.5 cm anterior to the ear at the tragus level. The needle will be inserted perpendicular to the skin and the fascia will be injected deeply and superficially while the needle is withdrawn. Postauricular branches of the greater auricular nerves will be blocked bilaterally with 2 ml of 0.5% bupivacaine injected 1 cm posterior to the ear, between the bone and skin, at the level of the tragus. The greater, lesser, and third occipital nerves run along the upper nuchal line approximately halfway between the occipital prominence and the mastoid prominence.
  Arms: scalp block
Other: Incisional infiltration — Incisional infiltration: 20 ml of 0.5% bupivacaine will be infiltrated by the surgeon into the PHHA points and surgical incision areas 10 minutes before PHHA. Two
  Arms: incisional infiltration

SUMMARY:
Postoperative pain after craniotomy is an important clinical problem as it can lead to hypertension and increased intracranial pressure. Multimodal analgesia methods are performed by anesthesiologists in different ways depending on the anesthetist's preference.

In addition, both techniques have been shown in studies to provide intraoperative hemodynamic stabilization in addition to their effects on postoperative pain. Although there are many studies on both techniques, the number of studies comparing scalp block with infiltration technique is very limited. Therefore, postoperative use of scalp block and incisional infiltration for postoperative pain after craniotomy is recommended.

DETAILED DESCRIPTION:
intraoperative Routine anesthesia induction will be applied after routine monitoring in the operating room. Anesthesia will be induced with propofol (1.5-2 mg/kg), rocuronium (0.6 mg/kg), fentanyl (1mcg/kg), 0.7 FiO2 oxygen. After intubation, general anesthesia will be maintained with the effect site model of target control infusion with propofol and remifentanil. Target concentrations will be maintained at 2 to 3 µg/ml propofol and 2 to 6 ng/ml remifentanil. The propofol dose was titrated according to the depth of anesthesia. The bispectral index will be kept between 45 and 60. Radial artery and urinary catheter will be inserted.

Group S: Following induction of anesthesia, a scalp block will be performed before the surgery begins.

Group I: Incisional infiltration will be performed before the surgery begins, following induction of anesthesia for the patient.

Scalp block: Scalp block will be performed by the anesthesiologist 10 minutes before the pin head holder application (PHHA). Supraorbital and supratrochlear nerves will be blocked bilaterally with 6 ml of 0.5% bupivacaine injected vertically into the skin above the eyebrow midline. Auriculotemporal nerves will be blocked bilaterally by injecting 4 ml of 0.5% bupivacaine 1.5 cm anterior to the ear at the tragus level. The needle will be inserted perpendicular to the skin and the fascia will be injected deeply and superficially while the needle is withdrawn. Postauricular branches of the greater auricular nerves will be blocked bilaterally with 2 ml of 0.5% bupivacaine injected 1 cm posterior to the ear, between the bone and skin, at the level of the tragus. The greater, lesser, and third occipital nerves will be blocked bilaterally with 8 ml of 0.5% bupivacaine injected along the upper nuchal line, approximately halfway between the occipital protuberance and the mastoid prominence.

Incisional infiltration: 20 ml of 0.5% bupivacaine will be infiltrated by the surgeon into the PHHA points and surgical incision areas 10 minutes before PHHA. If the mean arterial pressure (MAP) and heart rate increase above 20% of the baseline values in both groups, additional remifentanil 50 µg IV will be administered.

Intraoperative analgesia will be provided only with remifentanil. Sugammadex (2 mg/kg will be used to reverse the remaining muscle relaxation at the end of the surgery). Ondansetron (8 mg IV) will be administered as antiemetic prophylaxis. All patients will be extubated at the end of the surgery and will be admitted to the neurosurgery intensive care unit for 24 hours postoperatively.

Postoperative The per-operative analgesia plan will be applied the same to all patients. In this protocol, intravenous paracetamol 1 g. and tramadol was determined as 1mg/kg. Then it is paracetamol every eight hours and tramadol from PCA.

At the end of the operation, patients' pain levels will be determined and recorded using the Numeric Rating Scale (NRS) system at intervals in the first 24 hours postoperatively. NRS; It is a pain intensity determination system based on the system of having the person say a point between 0 (no pain), 10 (unbearable pain) and 10 (unbearable pain) to describe his/her pain. During service follow-ups, if NRS is 4 or above, 75 mg diclofenac sodium will be administered intramuscularly. Analgesia consumption amount, rescue analgesic needs and hours will be noted in detail, and rescue analgesic use as well as NRS scores at specified hours will be evaluated statistically. The postoperative analgesia plan will be applied the same to all patients. This protocol is our routine analgesia protocol that we apply in our hospital for cranial surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent craniotomy under elective conditions
2. ASA I-III
3. 18-75 years old
4. GCS >13

Exclusion Criteria:

1. GCS <13
2. Emergency surgery
3. Presence of contraindications to the LA agents used in this study
4. Chronic use of opioids
5. Psychiatric disorders
6. Presence of infection at the injection site
7. Uncontrolled intracranial hypertension
8. Chronic hypertension,
9. Coronary artery disease, arrhythmia,
10. Coagulopathy,
11. Patients who have previously undergone craniotomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 24 hours
  Postoperative 30th minute, 1st, 6th, 12th, 18th. Patients' opioid consumption on the PCA will be recorded at the 24th and 24th hours.

SECONDARY OUTCOMES:
The Numeric Rating Scale (NRS) | 24 hours
  Preoperative period and Postoperative 30th minute, 1st, 6th, 12th, 18th. And at the 24th hour, patients' pain levels and NRS scores will be recorded. At the end of the operation, patients' pain levels will be determined and recorded using the Numeric Rating Scale (NRS) system at intervals in the first 24 hours postoperatively. NRS; It is a pain intensity determination system based on the system of having the person say a point between 0 (no pain), 10 (unbearable pain) and 10 (unbearable pain) to describe his/her pain.

CONTACTS AND LOCATIONS:
Overall Officials: ferdi gülasştı, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Ferdi Gülaştı, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided